CLINICAL TRIAL: NCT06464432
Title: Complex-Posttraumatic Stress Disorder in Urban Egypt: Pilot Testing of a Culturally-adapted Evidence-Based Treatment Manual and Development of a Culture-specific Diagnostic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: The American University in Cairo (Other)
Responsible Party: Principal Investigator, Nadine Hosny, Doctoral Assistant, PhD Candidate, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 052024_00001; 2023-2024-204 (Other: American University in Cairo)
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Complex Post-Traumatic Stress Disorder

STUDY DESIGN:
Intervention Model Description: Un-randomized Pilot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: ESTAIR Psychotherapeutic Manual (Experimental)
  Interventions: Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation

INTERVENTIONS:
Behavioral: Enhanced Skills Training in Affective and Interpersonal Regulation — Enhanced Skills Training in Affective and Interpersonal Regulation combined with Modified Prolonged Exposure (ESTAIR); Psychotherapeutic manual for the treatment of Complex Post-Traumatic Stress Disorder (CPTSD) consisting of 4 therapeutic modules: 1. Emotion Regulation, 2, Self-concept, 3. Relationship Patterns, 4. Prolonged Exposure.

SUMMARY:
Background: The CPTSD diagnosis presented in the ICD-11 is supposed to provide core and culturally invariant symptoms, which is supported by recent research. Yet, evidence also shows the necessity of integrating culture-specific symptoms in intervention and diagnostic tools to enhance the validity and efficacy of such diagnoses and therapeutic interventions. Along with cultural aspects, there are relevant structural aspects e.g., economic, and social inequalities, which impact mental health. These aspects remain understudied in low middle income countries like Egypt, where there are considerable rates of violence.

Aims: The project aims to i) culturally adapt and pilot test the therapeutic manual ESTAIR/MPE in urban Egypt, and ii) to pilot test a cultural and structural module for the diagnostic assessment of CPTSD among the same target population. The objective is to assess the feasibility, acceptability, and initial impact on clinical outcomes of both the manual and diagnostic modules.

Methods: In earlier phases, the project gathered qualitative data from key informants on the cultural and structural dimensions of CPTSD in urban Egypt. Using the collected data, investigators culturally adapted this intervention and developed a diagnostic cultural module. Subsequently, the investigators will pilot-test it in four groups of five participants each, 20 participants in total. The project intends to collect both quantitative and qualitative measures to explore determined outcomes and analyze them accordingly.

DETAILED DESCRIPTION:
For further information, please see the attached protocol.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian
* 18 years of age or older
* Literate, can give written or oral consent
* History of severe and/or prolonged trauma, and screen positive for CPTSD
* Reside in any other major city

Exclusion Criteria:

* Imminent risk of suicide, psychotic symptoms, and/or severe alcohol and/or drug abuse
* Have been in therapy before (i.e., completed more than 5-10 sessions of psychotherapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility ESTAIR Manual | 7 months
  We will primarily assess feasibility by determining the percentage of participants who complete the study until the end (among those who sign the informed consent). Based on reported dropout rates from studies using similar modular interventions with trauma survivors, we will consider 80-90% participation and adherence as excellent, 70-80% as satisfactory, and 60-70% as acceptable.
Acceptability ESTAIR Manual | 7 months
  We will assess the acceptability by conducting feedback qualitative interviews after each module and overall feedback on therapy process at the end of therapy.
Feasibility of ITI-Cultural Module | 7 months
  We will assess the ITI feasibility, using the same method based on the percentage of participants who complete the ITI; 80-90% participation and adherence is considered as excellent, 70-80% as satisfactory, and 60-70% as acceptable.
Acceptability of ITI-Cultural Module | 7 months
  We will assess the acceptability of the ITI through qualitative interviews after the diagnostic interview.

SECONDARY OUTCOMES:
Complex post-traumatic stress disorder | 7 months
  The International Trauma Questionnaire asses 12 symptoms (6 for post-traumatic stress disorder and another 6 for disturbances in self-organisation). A diagnosis of CPTSD requires the endorsement of at least one of the two symptoms from each of the three PTSD symptom clusters described above (i.e., re-experiencing in the here and now, avoidance, and sense of current threat) and at least one of the two symptoms from each of the three Disturbances in Self-Organisation (DSO) clusters (i.e. affective dysregulation, negative self-concept, and disturbances in relationships). Items are scored on a Likert scale ranging from 0 (not at all) to 4 (extremely).
  The endorsement of a symptom item is defined as a score ≥ 2.
Depression | 7 months
  Patient Health Questionnaire (PHQ-9). The PHQ-9 score may range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of depression.
Anxiety | 7 months
  General Anxiety Disorder Questionnaire (GAD-7). The GAD-7 score may range from 0 to 21, since each of the 7 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores mean higher levels of anxiety.
Somatic Symptoms | 7 months
  Somatic Symptoms Scale (SSS-8). The SSS-8 score may range from 0 to 32, since each of the 8 items can be scored from 0 (not at all) to 4 (severely). Higher scores mean higher levels of somatic symptoms.
Well-being | 7 months
  WHO-5 questionnaire. Scores range from 0-25, based on a Likert scale from 0 (not at all) to 5 (all of the time) for each item. Higher scores reflect better levels of well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- The American University in Cairo, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT06464432/Prot_SAP_000.pdf